CLINICAL TRIAL: NCT03636776
Title: Prospective Study to Assess Quality of Life and Psychological Vulnerability in Patients With Metastatic Breast Cancer RH+
Brief Title: Quality of Life and Psychological Vulnerability in Patients With RH+ Metastatic Breast Cancer
Acronym: EPOCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor has set up a secondary competitive study concerning the same population and whose secondary objectives are the same as those of the EPOCA study with the same endpoints.
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-N-2015-04
Record Dates: First submitted 2018-08-08; First posted 2018-08-17 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Breast Cancer; Positive Hormonal Receptors
Keywords: Quality of Life; Psychological vulnerability
MeSH Terms: conditions — Breast Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- quality of life in metastatic BC (Experimental): Patients benefit from a longitudinal follow-up determined according to the treatments.
  Each type of treatment has its own schedule based on medical consultation times. At each change of treatment, from chemotherapy to hormone therapy or vice versa, the assessment times are determined according to the nature of the treatment.
  The rhythm of the evaluation visits will therefore be defined by the doctor, according to the habits of the centre.
  The evaluation times used to collect the questionnaires (QLQ-C30, BR23, PDS, STAI, BDI II).
  Interventions: Other: Quality of life in metastatic BC

INTERVENTIONS:
Other: Quality of life in metastatic BC — 1 month after metastatic stage diagnosis, patients complete their 1st therapeutic sequence evaluation visit (T1) within the recommended standard time frames. If the disease remains stable or if a response to treatment is observed then patients continue their follow-up in the same therapeutic sequence (T1).
  If progression occurs, treatment is modified and patients move on to the next therapeutic sequence (T2).
  And so on as many times as necessary. Before each evaluation visit with investigator, patients complete the questionnaires QLQ-C30, BR23, STAI, BDI II

SUMMARY:
Metastatic breast cancer (MBC) is a dark prognostic disease with survival at 5 years of less than 20% and a median survival of 24 to 30 months after diagnosis of metastasis. Thus, metastatic diagnosis can be expected to have a different impact on the quality of life of patients in early and advanced stages.

However, MBC benefits from therapeutics that improve patients' quality of life and even improve overall survival. The main objectives of this prospective study are :

* to evaluate the evolution over time of the quality of life of patients treated for positive hormonal receptors (RH+) metastatic breast cancer, according to the therapeutic class ;
* to evaluate the psychological vulnerability of these patients since the announcement of their metastatic diagnosis and during their treatments. Finally, when interviewing oncologists, to know the factors involved in a treatment change decision process for the same patient.

DETAILED DESCRIPTION:
Studying quality of life over time in patients followed for metastatic breast cancer will identify when a person may feel most vulnerable in their experience of the disease and treatment. A specific and adapted support can thus be set up throughout the disease, from the diagnosis and during the different phases of treatment.

Patients will benefit from a longitudinal follow-up determined according to the treatments. For example :

Chemotherapy : After the first assessment time at 1 month from diagnosis, patients receiving chemotherapy treatment are seen every 3 months.

Hormone therapy : After the first assessment time at 1 month from diagnosis, patients receiving hormone therapy are seen every 2 months.

Each type of treatment has its own schedule based on medical consultation times. At each change of treatment, from chemotherapy to hormone therapy or vice versa, the assessment times are determined according to the nature of the treatment.

The rhythm of the evaluation visits will therefore be defined by the doctor, according to the habits of the centre.

Patients will complete an end of study visit 3 years after inclusion

Quality of Life and Psychological vulnerability will be assessed through questionnaires :

* QLQ-C30 explores 5 functional scales (physical, social, psychological, cognitive functioning, daily activities) and 1 scale of health status and overall quality of life. It allows a detailed analysis of symptoms related to the disease and its treatment (fatigue, nausea/vomiting, pain, dyspnea, loss of appetite, sleep disturbance, constipation and diarrhea) as well as the financial impact for the patient.
* BR23 : specific questionnaire for breast cancer validated in French
* Psychological distress scale (PDS)
* State Trait Anxiety Inventory (STAI) : Assesses the feelings of apprehension, tension, nervousness and worry that the subject feels at the time of the anxiogenic or endangerment situation. This questionnaire is therefore an indicator of transient changes in anxiety caused by aversive or therapeutic situations.
* Beck Depression Inventory (BDI II) : assesses the severity of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of invasive breast cancer (=infiltrant). NB: Mixed histologies are allowed
2. Adult women (≥ 18 years),
3. Positive hormonal receptors (Estrogen receptors and/or Progesterone receptors ≥10%) and HER2 negative
4. Patient in need of a 1st metastatic treatment line NB: Patients may have received prior treatment for their cancer, but not for their metastatic disease.
5. Performance status ≤ 1 (world health organization)
6. Patients affiliated to a Social Security,
7. Obtaining the patient's signed written consent

Exclusion Criteria:

1. Patient with non-metastatic breast cancer,
2. man
3. Negative hormonal receptors or HER2 positive
4. Psychiatric history with specialist diagnosis
5. Pregnant or nursing patient
6. Patients who cannot be followed regularly for psychological reasons (cognitive problems preventing completion of questionnaires), or because of geographical remoteness.
7. Person deprived of liberty or adult under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline quality of life during breast cancer treatment | 3 years
  quality of life assessed using QLQ-C30 Questionnaire
Change from baseline psychological vulnerability during breast cancer treatment | 3 years
  Psychological vulnerability assessed using STAI questionnaire
Change from baseline quality of life during breast cancer treatment | 3 years
  quality of life assessed using BR23 Questionnaire
Change from baseline psychological vulnerability during breast cancer treatment | 3 years
  Psychological vulnerability assessed using Psychological distress scale. The scale represents a means of assessing the psychological state of patients. The scale measures 10 cm. The patients will have to put a cross on the line at the place which corresponds best to their psychological state of the past week. 0 indicates no distress and 10 very important distress.
Change from baseline psychological vulnerability during breast cancer treatment | 3 years
  Psychological vulnerability assessed using BDI-II questionnaire

SECONDARY OUTCOMES:
number of therapeutic class treatment prescribed during breast cancer treatment | 3 years
  The therapeutic strategy is modified in case of progression: chemotherapy and/or hormonotherapy. This change in treatment can affect the quality of life and psychological vulnerability of patients. The number of therapeutic classes prescribed in this way will make it possible to describe their impact over time on patients' quality of life and psychological vulnerability.

CONTACTS AND LOCATIONS:
Overall Officials: MARIO CAMPONE, MD, Principal Investigator — ICO NANTES
Locations (2):
- France (2):
  - Ico Angers, Angers
  - Ico Nantes, Saint-Herblain